CLINICAL TRIAL: NCT01811927
Title: The Treatment of Coronary Artery Lesions Using the PRO-Kinetic Energy Cobalt-Chromium, Bare-Metal Stent (BIOHELIX-II)
Brief Title: The Treatment of Coronary Artery Lesions Using the PRO-Kinetic Energy Cobalt-Chromium, Bare-Metal Stent
Acronym: BIOHELIX-II
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Biotronik AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C1210
Record Dates: First submitted 2013-03-13; First posted 2013-03-15 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PRO-Kinetic Energy Stent (Experimental): PRO-Kinetic Energy Stent
  Interventions: Device: PRO-Kinetic Energy Stent

INTERVENTIONS:
Device: PRO-Kinetic Energy Stent — Bare-metal stent

SUMMARY:
The purpose of this study is to the assess the clinical performance of the BIOTRONIK PRO-Kinetic Energy stent in subjects with atherosclerotic disease of native coronary arteries.

ELIGIBILITY:
Inclusion Criteria:

* Age > or = 18 years
* Willingness to comply with study follow-up requirements
* Candidate for a PCI procedure
* Candidate for coronary artery bypass graft surgery
* Documented evidence of stable or unstable angina pectoris or positive functional ischemia study (e.g. exercise treadmill test, thallium stress test, SPECT, stress echocardiogram or cardiac CT)
* Written informed consent
* De novo or restenotic lesion in a native coronary artery; restenotic lesions must have been previously treated with only standard PTCA (treatment must be > 12 months prior to the index procedure)
* Target lesion must be in a major coronary artery (target vessel). The target vessel includes the entire territory of the left anterior descending artery, left circumflex artery or right coronary artery and any major side branch of the artery.
* A maximum of one target lesion and one non-target lesion may be treated per subject. The lesions must be located in separate coronary arteries, with treatment of the non-target lesion occurring first using commercially available therapy (with exception of brachytherapy).
* Lesions may be one solid lesion or a series of multiple, smaller lesions to be treated as one lesion
* Target lesion must be treatable with a single investigational stent; an additional stent may be used when treating a vessel dissection or another similar intra-procedure complication (use of investigational stent preferred)
* Angiographic evidence of ≥ 50% and < 100% stenosis (by operator visual estimate) with a TIMI flow > 1
* Target lesion length of ≤ 31 mm by operator visual estimate
* Target vessel reference diameter of 2.25 mm to 4.0 mm by operator visual estimate

Exclusion Criteria:

* Baseline LVEF of < 30%; LVEF may be measured and assessed by standard-of-care echocardiography procedures within 90 days of the index procedure or by a left ventriculogram prior to the index procedure (operator visual assessment)
* PCI in any vessel 30 days prior to the index procedure or planned for within 30 days after the index procedure
* Stroke or transient ischemic attack within the last 6 months prior to enrollment
* Intolerance to contrast agents that cannot be medically managed and/or intolerance to antiplatelet, anticoagulant or thrombolytic medications
* Refusal of blood transfusions
* Any other medical condition, that in the opinion of the investigator, poses an unacceptable risk for implant of a stent according to the study indications
* Pregnant, planning to become pregnant or nursing during the course of the study. Women of child-bearing potential must have a negative blood pregnancy (beta hCG) test. Female subjects who are surgically sterile or post-menopausal are exempt from having a pregnancy test.
* Known allergy to L-605 CoCr alloy (cobalt, chromium, tungsten and nickel) or amorphous silicon carbide
* Life expectancy of less than one year
* Participation in any other clinical investigational device or drug study. Subjects may be concurrently enrolled in a post-market study, as long as the post-market study device, drug or protocol does not interfere with the investigational treatment or protocol of this study.
* Documented diagnosis of an acute MI within 72 hours of the index procedure and an elevation of Troponin or CKMB above the URL (CKMB measurement is not required if CK is normal) at the time of the index procedure (99th percentile of the individual investigative site's normal reference population)

  - For subjects with stable angina and elevated Troponin, CKMB <99% URL is required
* ECG changes consistent with an acute MI within 72 hours of the index procedure. ECG changes consistent with an acute MI include:

  * > 1 mm ST segment elevation or depression in consecutive leads
  * New LBBB
  * Development of pathological Q-waves in two contiguous leads of the ECG
* Acute coronary syndrome with baseline Troponin > 99% URL
* INR ≥ 1.6
* Concomitant renal failure with serum creatinine level > 2.5 mg/dL
* Unresolved neutropenia (white blood cell count < 3,000 / SL), thrombocytopenia (platelet count < 100,000 / SL) or thrombocytosis (platelet count > 700,000 / SL)
* Unprotected left main CAD (> 50% diameter stenosis by operator visual estimate)
* Target vessel has been treated with any PCI procedure (e.g. PTCA, stent, cutting balloon, atherectomy, etc.) within 12 months prior to the index procedure
* Target lesion has been treated with a stent, cutting balloon or atherectomy any time prior to the index procedure or has been treated with PTCA within 12 months prior to the index procedure
* Target vessel treated with brachytherapy anytime prior to index procedure
* Planned PCI in the target vessel within 9 months after the index procedure
* Target vessel has a non-target lesion with a > 50% stenosis that requires treatment during the index procedure
* Lesions preventing distal perfusion (TIMI flow 0 and 1) prior to wire crossing
* Target lesion is in the left main coronary artery or within 2 mm of the origin of the left anterior descending artery or left circumflex artery by operator visual estimate
* Target lesion is located within a saphenous vein graft or arterial graft
* Target lesion involves a bifurcation - lesion is located in a major coronary artery and involves a side branch with a diameter > 2 mm (by operator visual estimate)
* Presence of a complication following pre-dilatation of target lesion
* Presence of a complication following treatment of a non-target lesion (if applicable)
* Presence of a target vessel/lesion that has excessive tortuousity/angulation or is severely calcified preventing complete inflation of an angioplasty balloon
* Angiographic evidence of thrombus within the target lesion
* Target lesion is located within an aneurysm or associated with an aneurysm in the vessel segment either proximal or distal to the target lesion
* Use of cutting balloons, atherectomy or ablative devices immediately prior to investigational stent placement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2013-03; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
In-stent late lumen loss | 9-months post procedure

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Kaiser, Prof, Principal Investigator — University Hospital of Basel
Locations (3):
- St. Antonius Hospital, Nieuwegein, Netherlands
- Switzerland (2):
  - University Hospital of Basel, Basel
  - Kantonsspital St. Gallen, Sankt Gallen